CLINICAL TRIAL: NCT06782477
Title: A First-in-Human, Phase 1a, Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled, Single Ascending Dose Trial to Assess the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of STAR-0310 in Healthy Adult Participants
Brief Title: A Study of STAR-0310 in Healthy Adult Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Astria Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STAR-0310-101
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- STAR-0310 Dose 1 (Experimental): Participants will be randomized to receive STAR-0310 or matching placebo
  Interventions: Drug: STAR-0310; Drug: Placebo
- STAR-0310 Dose 2 (Experimental): Participants will be randomized to receive STAR-0310 or matching placebo
  Interventions: Drug: STAR-0310; Drug: Placebo
- STAR-0310 Dose 3 (Experimental): Participants will be randomized to receive STAR-0310 or matching placebo
  Interventions: Drug: STAR-0310; Drug: Placebo
- STAR-0310 Dose 4 (Experimental): Participants will be randomized to receive STAR-0310 or matching placebo
  Interventions: Drug: STAR-0310; Drug: Placebo
- STAR-0310 in Participants of Japanese Descent (Experimental): Participants will be randomized to receive STAR-0310 or matching placebo
  Interventions: Drug: STAR-0310; Drug: Placebo

INTERVENTIONS:
Drug: STAR-0310 — STAR-0310 will be administered as a subcutaneous bolus injection.
Drug: Placebo — Placebo will be administered as a subcutaneous bolus injection.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose trial evaluating the safety, tolerability, PK, and immunogenicity of STAR-0310 in healthy adult participants. There are 4 planned cohorts and potentially up to 1 additional cohort which may comprise of healthy adult participants of Japanese descent.

ELIGIBILITY:
Inclusion Criteria:

* Good health as determined by the Investigator based upon a medical evaluation.
* Body mass index (BMI) of 18 to 35 kg/m2 with a weight of at least 60 kg for men and at least 50 kg for women, with a maximum weight of 130 kg for any participant.
* Participants of childbearing potential must have a negative serum pregnancy test at Screening, agree to use highly effective forms of contraception and abstain from egg donation or fertility treatment
* Participants capable of producing sperm must use an effective method of contraception and abstain from sperm donation
* Healthy adults of Japanese descent, where both biological parents and all 4 biological grandparents are of Japanese ethnicity (applicable only for potential cohort of participants of Japanese descent).

Exclusion Criteria:

* Prior or ongoing medical condition that, in the Investigator's opinion, could adversely affect the safety of the participant.
* Known sensitivity to the ingredients of STAR-0310
* Taking any prescription or non-prescription medications within at least 5 half-lives or 7 days, whichever is longer, before the time of admission
* History of exposure to any biologic medication within 90 days or 5 half-lives, whichever is longer, before the time of admission
* Participation in a clinical trial involving receipt of an investigational product within 30 days (small molecule) or 90 days (biologics), or 5 half-lives, whichever is longer, before the time of admission

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events | [Time Frame: Day 1 through Day 252]

SECONDARY OUTCOMES:
Serum Concentration of STAR-0310 | [Time Frame: Day 1 (predose up to 2 hours before study drug administration, and 12 hours post dose), Days 2, 3, 7, 10, 14, 21, 28, 42, 56, 84, 112, 140, 168, 196, 224, 252 ]
  Blood samples will be collected to measure the serum concentration of STAR-0310 before and after study drug administration.
Number of Participants with Anti-drug Antibodies to STAR-0310 | [Time Frame: Day 1 predose, Days 14, 28, 84, 168, 252 ]
  Blood samples will be collected to assess the formation of STAR-0310 anti-drug antibodies in serum before and after study drug administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Austin Clinical Research Unit - Early Clinical Development, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No